CLINICAL TRIAL: NCT06675760
Title: The Effect of Mobile Augmented Reality Application on Nursing Students' Knowledge Skills and Motivation Regarding the Prevention and Assessment of Pressure Injuries
Brief Title: The Effect of Mobile Augmented Reality Application on Nursing Students' Knowledge Skills and Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Collaborators: Health Institutes of Turkey (Other Government); Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Emine SEZGÜNSAY, Lecturer, PhD Student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TUSEB-2022-ACIL-11-31345
Record Dates: First submitted 2024-10-30; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Education; Nursing
Keywords: nursing; Pressure Injury; augmented reality
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: : The research is a randomized controlled, quasi-experimental study. The population of the study consisted of 130 first-year students enrolled at Gülhane Faculty of Nursing, University of Health Sciences. Students were randomized into intervention and control groups using a computer program. A mobile augmented reality application was utilized to train students in the intervention group on pressure injury prevention, while students in the control group received traditional educational methods. Data collection occurred in two phases: preparation and implementation. In the preparation phase, presentation materials for the training, the mobile augmented reality application, and data collection forms were developed, and a pilot study was conducted. In the implementation phase, all students received the theoretical training together, while the laboratory sessions were conducted separately for each group. Then, the same evaluation steps were applied to all students.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the control groups (No Intervention): The control group received pressure injury assessment training through traditional education methods.
- The mobile augumented reality application intervention group (Experimental): The intervention group received training through a mobile augmented reality application in the laboratory.
  Interventions: Device: The intervention group

INTERVENTIONS:
Device: The intervention group — The intervention group received training through a mobile augmented reality application in the laboratory.
  Arms: The mobile augumented reality application intervention group

SUMMARY:
The aim of this study was to examine the effects of a mobile augmented reality application on nursing students' knowledge, skills, and motivation regarding pressure injuries.

DETAILED DESCRIPTION:
The research is a randomized controlled, quasi-experimental study. The population of the study consisted of 130 first-year students enrolled at Gülhane Faculty of Nursing, University of Health Sciences. In the study, a mobile augmented reality application was used for the training of students in the intervention group regarding pressure injury prevention. The training of the control group students continued with traditional education methods. The data collection process of the study was carried out in two stages: preparation and implementation. Prior to the commencement of the study, ethical committee approval and institutional permissions were obtained. In the analysis of the data, descriptive statistical methods such as number, percentage, min-max values, median, mean, and standard deviation were used, along with independent t-test, dependent t-test, and Chi-square analysis.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study.
* Taking the Fundamentals of Nursing course for the first time.

Exclusion Criteria:

* Using a language other than Turkish as a native language.
* Graduating from a Vocational Health High School.
* Being enrolled in the nursing faculty through vertical transfer.
* Working as a nurse or healthcare staff in a hospital or any healthcare institution.
* Being excluded from the control and experimental groups during randomization.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Student's knowledge scores | It used for first week of the research as a pre-test and fifth week of the research as a post-test
  The Pressure Ulcer Knowledge Assessment Tool (PUKAT 2.0), which assesses knowledge levels, was used to measure the study's primary outcome. Developed in 2017, this tool has a maximum score of 24, with higher scores indicating a greater level of knowledge (Manderlier et al., 2017).
Student's performance scores | It used fifth week of the research during the laboratory exam
  The Pressure Injury Evaluation Skill Checklist was used to evaluate student's performance scores. It was developed by the researcher based on expert feedback and was used to evaluate students' skills. Scores on the Pressure Injury Evaluation Skill Checklist range from 0 to 100, with higher scores indicating better performance in pressure injury skills.
Student's motivation scores | It used for first week of the research after the laboratory training
  The ARCS Motivation Learning Scale was used to measure student motivation scores. It was developed by Keller in 2010 (Keller, 2010). This scale has a scoring range of 0 to 165, with higher scores showing increased student motivation toward the course.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Gulhane Faculty of Nursing, Ankara, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manderlier B, Van Damme N, Vanderwee K, Verhaeghe S, Van Hecke A, Beeckman D. Development and psychometric validation of PUKAT 2.0, a knowledge assessment tool for pressure ulcer prevention. Int Wound J. 2017 Dec;14(6):1041-1051. doi: 10.1111/iwj.12758. Epub 2017 May 26. PMID 28547752